CLINICAL TRIAL: NCT02026011
Title: Optimizing Naltrexone for Individuals of East Asian Descent
Brief Title: Naltrexone for Individuals of East Asian Descent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NTX-AA; R01AA021744 (NIH)
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; naltrexone; Asian American; pharmacogenetics; OPRM1 gene
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; vivitrol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): Naltrexone 50 mg/day
  Interventions: Drug: Naltrexone
- Sugar pill (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Naltrexone is an opioid receptor antagonist with highest affinity for mu opioid receptors
  Other Names: Revia; Depade; Vivitrol
  Arms: Naltrexone
Drug: Placebo — Sugar pill, matched to the active study medication in capsule size and color
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
This study will elucidate the pharmacogenetic effects of the Asn40Asp SNP of the OPRM1 gene on biobehavioral and neural markers of response to naltrexone in individuals of East Asian descent, an ethnic group most likely to express the positive predictive allele.

DETAILED DESCRIPTION:
Recent pharmacogenetic studies have advanced the gene coding for µ-opioid receptors (OPRM1) gene as a potential moderator of responses to naltrexone. The most widely studied polymorphism of the OPRM1 gene is the Asn40Asp single nucleotide polymorphism (SNP), a functional mutation thought to affect receptor activity such that the Asp40 variant binds β-endorphin three times stronger than the Asn40 allele. Recent studies have found that Asp40 carriers have a stronger striatal dopamine response to intravenous alcohol administration and report stronger feelings of alcohol reward. Findings from the COMBINE Study demonstrated that if treated with Medication Management alone and naltrexone, 87.1% of Asp40 carriers had a good clinical outcome, compared with only 54.8% of Asn40 homozygotes. While these findings are promising, studies have also highlighted allele frequency imbalance as a function of ethnicity such that the Asp40 allele frequency is approximately 20% in Caucasians, 5% in individuals of African Ancestry, and as high as 50% among individuals of East Asian descent. Therefore, to the extent to which this SNP moderates behavioral and clinical responses to NTX, ethnicity must be carefully considered in order to extend the findings from primarily Caucasian samples to ethnic minorities, such as Asian Americans. Preliminary work by our team has found that among individuals of East Asian descent, Asp40 carriers show greater NTX-induced blunting of alcohol craving as well as potentiation of the aversive effects of alcohol. This pilot study also found support for a gene dose-response, such that Asp40Asp individuals showed greater NTX responsivity than those with the Asn40Asp genotype. This study seeks to build upon these preliminary findings by testing heavy drinkers of East Asian descent across three OPRM1 genotypes (Asn40Asn, n = 30; Asn40Asp, n = 30, and Asp40Asp, n = 30). Participants will complete two double-blinded, counterbalanced alcohol infusion and self-administration sessions, one after taking NTX (50 mg/day) and one after taking matched placebo for five days. In each medication condition, participants will complete a functional neuroimaging task examining cue-induced craving for alcohol. This study will elucidate the pharmacogenetic effects of the Asn40Asp SNP of the OPRM1 gene on biobehavioral and neural markers of response to naltrexone in individuals of Asian descent, an ethnic group most likely to express the positive predictive allele (Asp40). The long-term objective of this research is to optimize alcoholism pharmacotherapy and to address health disparities by advancing pharmacogenetic studies in ethnic minority groups.

ELIGIBILITY:
Inclusion Criteria:

* current (i.e., past month) alcohol dependence
* East Asian ethnicity (i.e., Chinese, Korean, or Japanese)
* Prospective genotyping for the A118G SNP of the mu opioid receptor (OPRM1) gene to allow for balanced groups on all three genotypes (AA, AG, GG)

Exclusion Criteria:

* lifetime DSM-IV of drug dependence (other than alcohol or nicotine)
* current use of psychoactive drugs as determined by self-reports and verified using toxicology testing
* lifetime diagnosis of bipolar disorder or any psychotic disorder
* contraindications to an MRI scan (including left handedness)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ray LA, Bujarski S, Chin PF, Miotto K. Pharmacogenetics of naltrexone in asian americans: a randomized placebo-controlled laboratory study. Neuropsychopharmacology. 2012 Jan;37(2):445-55. doi: 10.1038/npp.2011.192. Epub 2011 Sep 7. PMID 21900886
- See also: UCLA Addictions Laboratory — http://addictions.psych.ucla.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 199 individuals were screened in the laboratory, of those 106 completed the physical exam, and of those 87 were eligible and agreed to be randomized. Participants received in random order either Naltrexone (titrated up to 50 mg/day) or Placebo at each Allocation.
Groups:
- Allocated to Naltrexone: Group that was randomly assigned to receive Naltrexone first.
- Allocated to Placebo: Group that was randomly assigned to receive Placebo first
Period: Allocation 1 (First Set of Medication)
Arm/Group | Allocated to Naltrexone | Allocated to Placebo
Started | 46 | 41
Completed | 38 | 39
Not Completed | 8 | 2
Not completed — Side Effects | 6 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Investigator Withdrawal | 1 | 0
Period: Allocation 2 (Second Set of Medication)
Arm/Group | Allocated to Naltrexone | Allocated to Placebo
Started | 38 | 37
Completed | 37 | 35
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Providing baseline data for the 77 individuals who completed at least one experimental session
Groups:
- Asn40Asn Genotype: Group that is homozygotes for the Asn40 allele
- Asn40asp/Asp40Asp Genotype: Group that is a carrier of the Asp40 allele
- Total: Total of all reporting groups
Arm/Group | Asn40Asn Genotype | Asn40asp/Asp40Asp Genotype | Total
Number analyzed (Participants) | 29 | 48 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.72 (7.57) | 25.69 (4.84) | 26.83 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 19 | 28
  Male | 20 | 29 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Chinese | 12 | 13 | 25
  Ethnicity: Japanese | 2 | 6 | 8
  Ethnicity: Korean | 11 | 24 | 35
  Ethnicity: Taiwanese | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 48 | 77
Alcohol Use Disorder Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorder Identification Test (AUDIT) developed by the World Health Organization. The AUDIT is a 10 item measure from which you can calculate a total score ranging from 0 to 40. Higher scores indicate more hazardous drinking. A score = or > than 8 indicates a hazardous drinking pattern.
  units on a scale | 16.14 (5.82) | 13.17 (4.83) | 14.29 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: Subjective Response - Craving for Alcohol
Description: Alcohol Urge Questionnaire (AUQ) is used to assess subjective experiences of craving for alcohol. It consists of 8 items, each rated on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). A summary score is used at each assessment time point. The AUQ was administered at baseline and three levels of breath alcohol concentration: 0.02 g/dl. 0.04, g/dl, and 0.06 g/dl.
Time Frame: The AUQ was administered across a period of approximately 1.5 hours.
Population: Participants who completed at least one experimental session.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Naltrexone - Asn40Asn: Group that was randomized to receive Naltrexone (50 mg/d) and is homozygote for the Asn40 allele.
- Naltrexone - Asn40Asp/Asp40Asp: Group that was randomized to receive Naltrexone (50mg/d) and carries at least one copy of the Asp40 allele.
- Placebo - Asn40Asn: The group that was randomized to receive placebo and is homozygote for the Asn40 allele.
- Placebo - Asn40Asp/Asp40Asp: Group that was randomized to receive Placebo and carries at least one copy of the Asp40 allele.
Arm/Group | Naltrexone - Asn40Asn | Naltrexone - Asn40Asp/Asp40Asp | Placebo - Asn40Asn | Placebo - Asn40Asp/Asp40Asp
Number analyzed (Participants) | 27 | 48 | 28 | 46
score on a scale
  BrAC = 0.02 g/dl | 1.7037 (0.9295) | 1.9965 (1.2862) | 2.1012 (1.2881) | 1.8478 (0.9812)
  BrAC = 0.04 g/dl | 1.9198 (1.1260) | 2.1319 (1.3024) | 2.3095 (1.4499) | 2.2645 (1.2311)
  BrAc = 0.06 g/dl | 2.0185 (1.3590) | 2.2014 (1.3430) | 2.3095 (1.4400) | 2.4891 (1.4595)
Statistical Analysis 1: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.39, Mixed Models Analysis — Medication effect: b = -0.15, SE = 0.17, t = -0.86, p = 0.39
Statistical Analysis 2: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.34, Mixed Models Analysis — Genotype effect: b = 0.20, SE = 0.21, t = 0.96, p = 0.34
Statistical Analysis 3: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — BrAC effect: b = 0.13, SE = 0.06, t = 2.10, p = 0.04
Statistical Analysis 4: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.47, Mixed Models Analysis — Medication by genotype interaction: b = 0.15, SE = 0.21, t = 0.73, p = 0.47
Statistical Analysis 5: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis — Medication by genotype by BrAC interaction: b = -0.20, SE = 0.13, t = -1.52, p = 0.13

2. Primary Outcome: Subjective Response - Stimulation
Description: The Biphasic Alcohol Effects Scale (BAES) Stimulant Subscale consists of 14 items designed to capture the stimulant effects of alcohol, rated on an 11-point scale (0 = not at all. 10 = extremely). Total score for the stimulant subscale ranges from 0-70.
Time Frame: The BAES Stimulant Subscale was administered at baseline and three levels of breath alcohol concentration: 0.2 g/dl. 0.04, g/dl, and 0.06 g/dl taking place within approximately 1.5 hours
Population: Participants who completed at least one experimental session.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo - Asn40Asn: The group that was randomized to receive placebo first and is homozygote for the Asn40 allele.
Arm/Group | Naltrexone - Asn40Asn | Naltrexone - Asn40Asp/Asp40Asp | Placebo - Asn40Asn | Placebo - Asn40Asp/Asp40Asp
Number analyzed (Participants) | 27 | 48 | 28 | 46
score on a scale
  BrAC = 0.02 g/dl | 2.0423 (1.7338) | 2.0893 (1.8291) | 2.0102 (1.9867) | 1.8106 (1.7512)
  BrAC = 0.04 g/dl | 2.2963 (1.8860) | 2.7679 (1.9415) | 2.3316 (2.0949) | 2.4658 (1.9971)
  BrAc = 0.06 g/dl | 2.8307 (2.3581) | 3.0149 (2.1955) | 2.2347 (1.9917) | 3.0466 (2.4146)
Statistical Analysis 1: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.23, Mixed Models Analysis — Medication effect: b = 0.16, SE = 0.13, t = 1.20, p = 0.23
Statistical Analysis 2: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis — Genotype effect: b = 0.37, SE = 0.22, t = 1.69, p = 0.09
Statistical Analysis 3: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis — Medication by genotype interaction: b = 0.04, SE = 0.21, t = 0.20, p = 0.84
Statistical Analysis 4: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis — Medication by genotype by BrAC interaction: b = -0.32, SE = 0.16, t = -1.93, p = 0.05

3. Primary Outcome: Subjective Response - Sedation
Description: The Biphasic Alcohol Effects Scale (BAES) Sedation Subscale consists of 14 items designed to capture the sedating effects of alcohol, rated on an 11-point scale (0 = not at all. 10 = extremely). Total score for the sedation subscale ranges from 0-70.
Time Frame: The BAES Sedation Subscale was administered at baseline and three levels of breath alcohol concentration: 0.2 g/dl. 0.04, g/dl, and 0.06 g/dl taking place within approximately 1.5 hours
Population: Participants who completed at least one experimental session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone - Asn40Asn | Naltrexone - Asn40Asp/Asp40Asp | Placebo - Asn40Asn | Placebo - Asn40Asp/Asp40Asp
Number analyzed (Participants) | 27 | 48 | 28 | 46
score on a scale
  BrAC = 0.02 g/dl | 2.6825 (2.1146) | 2.3482 (1.6194) | 2.1480 (1.6452) | 2.0560 (1.6726)
  BrAC = 0.04 g/dl | 2.8571 (2.1907) | 2.8601 (2.0094) | 2.4949 (1.7798) | 2.6832 (1.8504)
  BrAc = 0.06 g/dl | 3.0688 (2.4364) | 3.1548 (2.0981) | 2.6786 (2.4767) | 2.4627 (1.8025)
Statistical Analysis 1: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis — Medication effect: b = 0.14, SE = 0.23, t = 0.61, p = 0.55
Statistical Analysis 2: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis — Genotype effect: b = -0.11, SE = 0.37, t = -0.30, p = 0.77
Statistical Analysis 3: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — BrAC effect: b = 0.30, SE = 0.15, t = 2.02, p = 0.04
Statistical Analysis 4: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.47, Mixed Models Analysis — Medication by genotype interaction: b = -0.21, SE = 0.29, t = -0.72, p = 0.47
Statistical Analysis 5: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.19, Mixed Models Analysis — Medication by genotype by BrAC interaction: b = 0.28, SE = 0.21, t = 1.30, p = 0.19

4. Primary Outcome: Neural Response to Alcohol Cues
Description: Alcohol taste cues task for functional magnetic resonance imaging (fMRI). Region of Interest (ROI) were atomically defined using the Harvard-Oxford atlas in standard Montreal Neurological Institute (MNI) space, which were transformed into individual participants' native space using Functional Magnetic Resonance Imaging of the Brain Software Library (FSL). Contrast estimates are for Alc > Water cue, and are arbitrary units.
Time Frame: During the alcohol cue exposure fMRI paradigm which is expected to last 45 minutes
Population: Participants who completed at least one experimental session and whose neuroimaging data was not excluded due to excessive motion (>2 mm translation) and/or poor registration.
Measure: Mean (Standard Deviation); unit: Mean contrast estimate for Alc>Water cue
Arm/Group | Naltrexone - Asn40Asn | Naltrexone - Asn40Asp/Asp40Asp | Placebo - Asn40Asn | Placebo - Asn40Asp/Asp40Asp
Number analyzed (Participants) | 18 | 23 | 18 | 23
Mean contrast estimate for Alc>Water cue
  Ventral Striatum | 1.48 (19.94) | 8.07 (13.95) | .53 (13.47) | 1.03 (13.54)
  Orbitofrontal cortex | .12 (11.75) | 4.43 (9.64) | .45 (7.2) | 3.56 (6.95)
  Anterior Cingulate cortex | 3.31 (17.96) | 7.04 (13.90) | 5.17 (14.24) | 9.49 (13.07)

5. Secondary Outcome: Alcohol Self-administration - Number of Drinks
Description: Total number of drinks consumed during the alcohol self-administration task
Time Frame: Alcohol self-administration period was 1 hour long
Population: Participants who completed at least one experimental session.
Measure: Mean (Standard Deviation); unit: drinks consumed
Arm/Group | Naltrexone - Asn40Asn | Naltrexone - Asn40Asp/Asp40Asp | Placebo - Asn40Asn | Placebo - Asn40Asp/Asp40Asp
Number analyzed (Participants) | 27 | 48 | 28 | 46
drinks consumed | 1.4444 (1.5275) | 0.6458 (1.1576) | 1.5714 (1.4764) | 0.9565 (1.3656)
Statistical Analysis 1: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.14, Poisson Regression — Medication effect: F(1,71) = 2.24, p = 0.14
Statistical Analysis 2: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.02, Poisson — Genotype effect: F(1, 71) = 5.79, p = 0.02
Statistical Analysis 3: Comparison: Naltrexone - Asn40Asn vs Naltrexone - Asn40Asp/Asp40Asp vs Placebo - Asn40Asn vs Placebo - Asn40Asp/Asp40Asp; Test type: Superiority or Other; p = 0.41, Poisson — Medication by genotype interaction: F(1, 70) = 0.68, p = 0.41

ADVERSE EVENTS:
Time Frame: Adverse event data were collected immediately prior to alcohol infusion while on naltrexone and while on placebo (2 time points). This data was collected twice for each participant, once while they were on placebo and once while they were on naltrexone.
Description: Adverse events are defined as any symptom endorsed on the Side Effects Checklist (SAFTEE). The instructions on the SAFTEE are, "Have you noticed any of the following symptoms within the last 6 hours? If yes, how severe were the symptoms? Do you believe these symptoms were caused by the study medication?"
Arm/Group | Naltrexone | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/74
Other Adverse Events (participants affected / at risk) | 35/75 | 22/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=75) | Sugar Pill (N=74)
Abdominal pain or cramps (Gastrointestinal disorders) | 5 | 4
Yellow Eyes (Eye disorders) | 0 | 0
Nausea or vomiting (Gastrointestinal disorders) | 8 | 2
Irritability or anger (General disorders) | 7 | 0
Increased desire for sex (General disorders) | 4 | 3
Nervousness (General disorders) | 5 | 3
Ringing in the ears (General disorders) | 2 | 1
Decrease in appetite (General disorders) | 11 | 2
Depression (General disorders) | 2 | 1
Fatigue (General disorders) | 18 | 8
Difficulty in staying awake (General disorders) | 10 | 4
Increase in appetite (General disorders) | 3 | 3
Blurred vision (Eye disorders) | 3 | 0
Drowsiness (General disorders) | 15 | 5
Headache (General disorders) | 4 | 4
Night sweats (General disorders) | 1 | 2
Mental confusion (General disorders) | 3 | 1
Anxiety (General disorders) | 7 | 3
Joint or muscle pain (General disorders) | 2 | 1
Dizziness (General disorders) | 3 | 1
Sexual problems (General disorders) | 1 | 0
Difficulty sleeping (General disorders) | 8 | 6
Fever or chills (General disorders) | 1 | 1
Decreased desire for sex (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No